CLINICAL TRIAL: NCT00509262
Title: A Multicenter, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Sitagliptin Versus Glipizide in Patients With Type 2 Diabetes Mellitus and Chronic Renal Insufficiency Who Have Inadequate Glycemic Control
Brief Title: Sitagliptin Versus Glipizide in Participants With Type 2 Diabetes Mellitus and Chronic Renal Insufficiency (MK-0431-063 AM1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0431-063; 2007_549 (Other: Merck Registration Number)
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Results first posted 2012-03-28 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — Sitagliptin Phosphate; Glipizide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin + Placebo for Glipizide
  Interventions: Drug: Sitagliptin; Drug: Placebo for Glipizide
- Glipizide (Active Comparator): Glipizide + Placebo for Sitagliptin
  Interventions: Drug: Glipizide; Drug: Placebo for Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — Participants with moderate renal insufficiency will receive two sitagliptin 25 mg tablets orally daily; participants with severe renal insufficiency will receive one sitagliptin 25 mg tablet orally daily
  Other Names: MK-0431; Januvia
  Arms: Sitagliptin
Drug: Glipizide — Participants will receive glipizide 2.5 mg (1/2 tablet) orally once daily up to 20 mg orally daily (10 mg twice daily)
  Other Names: Glucotrol
  Arms: Glipizide
Drug: Placebo for Sitagliptin — Participants with moderate renal insufficiency will receive 2 placebo for sitagliptin tablets orally daily; participants with severe renal insufficiency will receive 1 placebo for sitagliptin tablet orally daily
  Arms: Glipizide
Drug: Placebo for Glipizide — Participants will receive 1/2 tablet of placebo for glipizide orally once daily up to 2 tablets orally twice daily
  Arms: Sitagliptin

SUMMARY:
The purpose of the study is to compare how sitagliptin and glipizide lower blood glucose levels in participants with moderate or severe renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes mellitus
* Has moderate or severe renal insufficiency

Exclusion Criteria:

* Has type 1 diabetes mellitus or a history of ketoacidosis
* Is on a new weight loss program
* Has active liver disease
* Is on dialysis or is likely to need dialysis during the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2007-10-09 (Actual); Primary Completion 2011-03-16 (Actual); Study Completion 2011-03-16 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Arjona Ferreira JC, Marre M, Barzilai N, Guo H, Golm GT, Sisk CM, Kaufman KD, Goldstein BJ. Efficacy and safety of sitagliptin versus glipizide in patients with type 2 diabetes and moderate-to-severe chronic renal insufficiency. Diabetes Care. 2013 May;36(5):1067-73. doi: 10.2337/dc12-1365. Epub 2012 Dec 17. PMID 23248197

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One site was identified as non-compliant with some of the requirements of Good Clinical Practice. For this reason, data from the 3 participants randomized at this site were deemed unreliable and were removed from all analyses.
Groups:
- Sitagliptin: Participants randomized to 25 or 50 mg of sitagliptin orally daily + placebo for glipizide
- Glipizide: Participants randomized to glipizide 2.5 to 20 mg orally daily + placebo for sitagliptin
Period: Overall Study
Arm/Group | Sitagliptin | Glipizide
Started | 211 | 212
Completed | 164 | 170
Not Completed | 47 | 42
Not completed — Adverse Event | 16 | 18
Not completed — Other | 2 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 6
Not completed — Physician Decision | 1 | 3
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 24 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Glipizide | Total
Number analyzed (Participants) | 211 | 212 | 423
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (10.7) | 64.2 (9.4) | 64.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 90 | 170
  Male | 131 | 122 | 253

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (A1C) Levels at Week 54
Description: A1C represents percentage of glycosylated hemoglobin.
Time Frame: Baseline to Week 54
Population: The per protocol population required that a participant had measurements both at baseline and at Week 54, and did not have any major protocol violations (e.g. drug compliance <75%, addition of prohibited antihyperglycemic agent, or incorrect double-blind study medication). No missing data were imputed.
Measure: Mean (Standard Deviation); unit: Percent of glycosylated hemoglobin
Groups:
- Sitagliptin: Participants received 25 or 50 mg of sitagliptin orally daily + placebo for glipizide
- Glipizide: Participants received glipizide 2.5 to 20 mg orally daily + placebo for sitagliptin
Arm/Group | Sitagliptin | Glipizide
Number analyzed (Participants) | 135 | 142
Percent of glycosylated hemoglobin
  Baseline | 7.76 (0.65) [-0.89 to -0.62] | 7.79 (0.70) [-0.64 to -0.51]
  Change from Baseline at Week 54 | -0.70 (0.80) | -0.62 (0.91)
Statistical Analysis 1: Comparison: Sitagliptin vs Glipizide; Test type: Non-Inferiority or Equivalence — The pre-specified non-inferiority margin was 0.4%; i.e., non-inferiority required that the upper boundary of the 95% confidence interval for the treatment difference (sitagliptin minus glipizide) to be less than 0.4%; ANCOVA; Difference in least squares mean = -0.11, 95% CI 2-sided [-0.29 to 0.06], Standard Deviation 0.74 — Based on analysis of covariance with terms for treatment, renal insufficiency stratum at Visit 4/Week -2 (moderate, or severe), prior diabetes pharmacotherapy (on or not on oral antihyperglycemic agent), and a covariate for baseline A1C

2. Primary Outcome: Percentage of Participants With Hypoglycemic Events
Description: Percentage of participants with at least one symptomatic hypoglycemic adverse event, excluding data after initiation of glycemic rescue therapy.
Time Frame: Baseline up to 28 days following the last dose of study therapy
Population: All participants as treated (APaT) population included all randomized participants who took at least one dose of study therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Sitagliptin | Glipizide
Number analyzed (Participants) | 210 | 212
percentage of participants | 6.2 | 17.0
Statistical Analysis 1: Comparison: Sitagliptin vs Glipizide; Test type: Superiority or Other; p = 0.001, Miettirnen& Nurminen method; Mean Difference (Final Values) = -10.8, 95% CI 2-sided [-17.1 to -4.8] — Miettirnen & Nurminen method stratified by renal insufficiency stratum at Visit 4/Week -2 (moderate or severe) & prior diabetes pharmacotherapy

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 54
Time Frame: Baseline to Week 54
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin | Glipizide
Number analyzed (Participants) | 136 | 142
mg/dL
  Baseline | 148.6 (39.9) | 143.9 (35.7)
  Change from Baseline at Week 54 | -16.7 (47.1) | -20.2 (48.6)
Statistical Analysis 1: Comparison: Sitagliptin vs Glipizide; Test type: Superiority or Other; ANCOVA; Difference in least squares mean = 7.1, 95% CI 2-sided [-1.9 to 16.1], Standard Deviation 38.3 — Analysis of covariance with terms for treatment, renal insufficiency stratum at Visit 4/Week -2 (moderate or severe), prior diabetes pharmacotherapy (on or not on oral antihyperglycemic agent), and a covariate for baseline Fasting Plasma Glucose

4. Secondary Outcome: Change From Baseline in Body Weight at Week 54
Time Frame: Baseline to Week 54
Population: All participants as treated (APaT) population included participants who had both baseline and Week 54 data (excluding data after initiation of glycemic rescue therapy).
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Sitagliptin | Glipizide
Number analyzed (Participants) | 143 | 148
kg | -0.6 (0.3) | 1.2 (0.3)
Statistical Analysis 1: Comparison: Sitagliptin vs Glipizide; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in least squares mean = -1.8, 95% CI 2-sided [-2.6 to -1.0], Standard Deviation 3.8 — Analysis of covariance with terms of treatment, renal insufficiency stratum at Visit 4/Week -2 (moderate or severe), prior diabetes pharmacotherapy (on or not on oral antihyperglycemic agent), and a covariate for baseline body weight

ADVERSE EVENTS:
Description: One participant from the sitagliptin group did not receive any study medication and, therefore, was excluded from all analyses. Analyses of safety used the APaT population (participants who had both baseline and Week 54 data, and for serious adverse events only, included data after the initiation of glycemic rescue therapy).
Arm/Group | Sitagliptin | Glipizide
Serious Adverse Events (participants affected / at risk) | 36/210 | 38/212
Other Adverse Events (participants affected / at risk) | 69/210 | 89/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=210) | Glipizide (N=212)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (3)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 3 (3)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Uraemic gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (3)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 2 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=210) | Glipizide (N=212)
Diarrhoea (Gastrointestinal disorders) | 11 (14) | 12 (13)
Oedema peripheral (General disorders) | 15 (17) | 10 (11)
Upper respiratory tract infection (Infections and infestations) | 10 (15) | 15 (19)
Urinary tract infection (Infections and infestations) | 11 (13) | 20 (31)
Blood glucose decreased (Investigations) | 15 (29) | 32 (159)
Hypoglycaemia (Metabolism and nutrition disorders) | 12 (21) | 35 (89)
Dizziness (Nervous system disorders) | 7 (7) | 11 (12)
Hypertension (Vascular disorders) | 11 (11) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.